CLINICAL TRIAL: NCT02253966
Title: Preoperative Intraarticular Injection of Methylprednisolone in Patients Scheduled for Total Knee-arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Iben Engelund Luna, MD, Research Fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-3-2014-089
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Knee Joint Osteoarthrosis; Hyperalgesia; Severe Movement Related Pain
MeSH Terms: conditions — Hyperalgesia | interventions — Methylprednisolone Acetate; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisoloneacetate (Active Comparator): Administration of:
  1 ml methylprednisoloneacetate 40 mg/ml 5 ml lidocaine 20 mg/ml 4 ml sodium chloride 9 mg/ml as a single intraarticular injection 7 days prior to surgery.
  Interventions: Drug: Methylprednisoloneacetate; Drug: Lidocaine; Other: sodium chloride
- Sodium chloride (Placebo Comparator): Administration of:
  5 ml lidocaine 20 mg/ml 5 ml sodium chloride 9 mg/ml as a singe intraarticular injection 7 days prior to surgery.
  Interventions: Drug: Lidocaine; Other: sodium chloride

INTERVENTIONS:
Drug: Methylprednisoloneacetate
  Other Names: Depo-Medrol
  Arms: Methylprednisoloneacetate
Drug: Lidocaine
Other: sodium chloride
  Other Names: saline

SUMMARY:
Despite improvements in analgesic treatment following total knee arthroplasty (TKA) for osteoarthrosis, a substantial part of patients still have severe acute pain after surgery. It has been suggested that preoperative degree of intraarticular inflammation is associated to postoperative degree of pain and level of function. Furthermore it is known, that patients with preoperative inflammation have hyperalgesia and severe movement related pain.

The aim of this study is to investigate the effect of a preoperative intraarticular injection of Methylprednisoloneacetate in reducing acute postoperative pain after total knee arthroplasty in patients with signs of severe pre-operative inflammation and pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 -80
* Osteoarthrosis
* Scheduled for primary unilateral TKA
* Preoperative pain report with NRS > 5 upon walking
* Signs of sensitisation in knee

Exclusion Criteria:

* Allergies to methylprednisoloneacetate, lidocaine or standard analgesic treatment
* Deficient written or spoken danish
* Impairment from psychological or neurological disease
* Local og systemic infection
* Immunodeficiency
* Treatment with corticosteroid within 30 days of inclusion
* Insulin treated diabetes mellitus
* Anticoagulant therapy
* ASA (American Society of Anaesthesia) class > 3
* General anaesthesia
* Alchohol use > 21 units / week
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours postoperatively
  Pain intensity on a numeric rang scale (NRS) from 0 to 10 upon ambulation 24 hours following surgery

SECONDARY OUTCOMES:
Pain | 48 hours postoperatively
  Pain intensity on a NRS from 0 to 10 upon ambulation 48 hours following
Pain | From day 1 to day 14
  Diary-reported pain intensity on a NRS from 0 to 10 when walking. Once daily from first to fourteenth postoperative day
Pain | From day 1 to day 14
  Diary-reported pain intensity on a NRS from 0 to 10 upon rest. Once daily from first to fourteenth postoperative day
Sensitisation | On day 0 and day 2
  Quantitative sensory testing (temporal summation / pressure algometry) on the day of surgery and on the second postoperative day.
Inflammation | On day 0 and day 2
  Measurement of C-reactive protein in blood sample on the day of surgery and on the second postoperative day.
Inflammation | On day 0
  Measurement of interleukin-6 level in knee joint fluid on the day of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark